CLINICAL TRIAL: NCT03833141
Title: Patient Outcomes Real World Evidence Registry (POWER): Patient Reported Outcomes in a Cohort of Canadian Adults With Severe Eosinophilic Asthma on Benralizumab.
Brief Title: Patient Reported Outcomes in Adults With Severe Eosinophilic Asthma on Benralizumab.
Acronym: POWER
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00041
Record Dates: First submitted 2018-10-11; First posted 2019-02-06 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Severe Eosinophilic Asthma
MeSH Terms: conditions — Pulmonary Eosinophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey Administration — Patient Reported Outcomes (PROs) of health, quality of life, and economic outcomes during routine clinical practice.
  Other Names: PRO survey

SUMMARY:
This study will generate patient reported outcomes (PROs) associated with the use of benralizumab as treatment for severe eosinophilic asthma.

DETAILED DESCRIPTION:
Benralizumab was launched in 2018 following regulatory approval in Canada and is now widely available for Canadian patients with severe eosinophilic asthma.

This study is an observational cohort study of patient reported outcomes (PROs) within real-world settings for participants who are prescribed benralizumab for treatment of uncontrolled severe eosinophilic asthma. Patients will be recruited in select clinics across Canada.

Survey data for each participant in the study will be obtained at the following time-points:

* Baseline (Week 0)
* Short-term follow up: 1-, 2-, 4-, and 8-weeks after baseline
* Long-term follow-up: 24- and 56-weeks after baseline

ELIGIBILITY:
The following individuals may be eligible to participate:

* Are enrolled in the benralizumab PSP;
* Are 18 years of age or older;
* Can understand the requirements of the study and provide informed consent to participate in this study;
* Agree to abide by the study protocol and the exclusion criteria and can complete all aspects of the study, including all visits.
* Are benralizumab naïve and have not previously received benralizumab prior to the start of this study

AND

* Suffer from uncontrolled severe eosinophilic asthma meeting at least one of the following:

  1. Has blood eosinophil count ≥ 300 cells/μL AND experienced two or more clinically-significant exacerbations in the past 12 months; OR
  2. Has blood eosinophil count ≥ 150 cells/μL AND are treated chronically with oral corticosteroids (OCS); OR
  3. Sputum eosinophil levels of 3% and higher OR
  4. Have been previously treated with a biologic for severe asthma and previously met the above eosinophil counts (detailed in #1,2, or 3 above) prior to initiation of the previous biologic.

     AND
* ACQ-6 score ≥ 1.5

Exclusion criteria:

Any of the following conditions are cause for exclusion from the study:

* Patients currently enrolled in an interventional clinical study in parallel will be excluded from the study, except for patients who are in parallel documented in a national asthma registry;
* Patients who have previously received benralizumab prior to the start of the study
* Patients currently participating (i.e. have not completed) in any other clinical trial including those with biologic treatment;
* Patients with other documented lung disease other than asthma and not within reimbursed label.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Canadian adults (18+) with uncontrolled severe eosinophilic asthma.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Change of at least 0.5 units in ACQ-6 after initiation of benralizumab | Up to week 56 (from 1st dose of benralizumab)
  ACQ-6 is able to identify the adequacy of asthma control in individual patients.
  Data will be presented as the proportion of patients achieving a change of at least 0.5 units following initiation of therapy.

SECONDARY OUTCOMES:
Number of exacerbations | Up to week 56 (from first dose of benralizumab)
  The start of an exacerbation is defined as the start-date of systemic corticosteroids or start-date of a temporary increase in a stable oral corticosteroid background dose, or start-date of a hospital admission, whichever occurs earlier.
  Data will be presented as an annualized exacerbation rate.
Change in concomitant medications | Up to week 56 (from first dose of benralizumab)
  Change in concomitant medications (i.e. oral corticosteroid usage) will be measured.
Number of participants with Serious Adverse Events and hospitalizations | Up to week 56 (from first dose of benralizumab)
  Assessment of safety and tolerability through measuring the overall change in number of serious adverse events and hospitalizations.
  Data will be presented as the proportion of patients experiencing serious adverse events and hospitalizations.
Asthma Quality of Life Questionnaire, Symptoms (AQLQ(S)+12) | Up to week 56 (from first dose of benralizumab)
  The AQLQ(S)+12 is a questionnaire that measures the health-related quality of life experienced by asthma patients.
  The questionnaire comprises 4 separate domains (symptoms, activity limitations, emotional function, and environmental stimuli).
  Patients are asked to recall their experiences during the previous 2 weeks and to score each of the questions on a 7-point scale ranging from 7 (no impairment) to 1 (severe impairment). The overall score is calculated as the mean response to all questions, and is presented as a score from 1 to 7, with lower overall scores indicating increasing impairement.
  The 4 individual domain scores (symptoms, activity limitations, emotional function, and environmental stimuli) are the means of the responses to the questions in each of the domains.
  Individual AQLQ(s)+12 Total or domain score changes of ≥0.5 are considered clinically meaningful.
  Data will be presented as a mean score and change from baseline with a measure of dispersion.
Health care resource utilization | Up to week 56 (from first dose of benralizumab)
  Health Care Resource Utilization (HCRU) will be measured through the overall change in the number of hospitalization visits, visits to the emergency department, and presenteeism/absenteeism from school/work.
EuroQol 5 Dimension, 5 Level (EQ-5D-5L) | Up to week 56 (from first dose of benralizumab)
  The EQ-5D-5L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The measurement of the EQ-5D-5L health states, defined by the EQ-5D-5L descriptive system, may be converted into a single index value. The index values, presented in country specific value sets, are a major feature of the EQ-5D instrument, facilitating the calculation of quality-adjusted life years (QALYs) that are used to inform economic evaluations of health care interventions.
  Index values are presented on a continuum between 0 and 1, with values approaching 1 indicating increasing quality of life (utility).
  Data will be presented as mean score as well as a change from baseline score with a measure of dispersion.
Treatment Satisfaction Questionnaire for Medication (TSQM-9) | Up to week 56 (from first dose of benralizumab)
  The TSQM-9 treatment satisfaction questionnaire is a measure of Effectiveness, Side effects, Convenience, and Global Satisfaction. The scores range from 0 to 100 with higher scores indicating greater satisfaction.
  Data will be presented as a mean score with a change from baseline calculation including a measure of dispersion.
Patient Global Impression of Change (PGIC) | Up to week 56 (from first dose of benralizumab)
  The self-reported measure Patient Global Impression of Change (PGIC) reflects a patient's belief about the efficacy of treatment.
  PGIC is a 7 point scale depicting a patient's rating of overall improvement.
  Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
  Data will be presented as a mean score with a change from baseline calculation including a measure of dispersion.
Patient Global Impression of Severity (PGI-S) | Up to week 56 (from first dose of benralizumab)
  PGI-S is a 1-item questionnaire designed to assess patient's impression of disease severity. The PGI-S item asks the participant to best describe how their asthma symptoms are now ("Check the one number that best describes how your asthma symptoms are now") on a 4-point scale scored as: "normal" (1), "mild" (2), "moderate" (3), or "severe" (4) .
  Data will be presented as a mean score with a change from baseline calculation including a measure of dispersion.

CONTACTS AND LOCATIONS:
Overall Officials: Erika Penz, MD, Principal Investigator — University of Saskatchewan
Locations (16):
- Canada (16):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Red Deer, Alberta
  - Research Site, Sherwood Park, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Bathurst, New Brunswick
  - Research Site, Ajax, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, North Bay, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Barrie, Ontaro
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Regina, Saskatchewan
  - Research Site, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No